CLINICAL TRIAL: NCT00794313
Title: Quantification of the Antidyskinetic Effect of Amantadine and Topiramate in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Ended
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kathryn Anne Chung, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: e4717
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinsons disease; dyskinesia; amantadine; efficacy
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Amantadine; Topiramate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amantadine (Experimental)
  Interventions: Drug: Amantadine 300 mg
- Amantadine plus Topiramate (Experimental)
  Interventions: Drug: Amantadine 300 mg; Drug: Topiramate
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Amantadine 300 mg — Amantadine, 300 mg, capsule, three times a day, two weeks
  Arms: Amantadine; Amantadine plus Topiramate
Drug: Topiramate — Topiramate, 25 mg, capsule, two times a day, 1 week Sugar Pill, capsule, one time a day, 1 week Topiramate, 50 mg, capsule, three times a day, 1 week
  Other Names: Topamax
  Arms: Amantadine plus Topiramate
Drug: Sugar Pill — sugar pill, capsule, three times a day, 2 weeks
  Arms: Sugar Pill

SUMMARY:
Levodopa is the main drug treatment for Parkinson's disease. Levodopa can cause unwanted and uncontrolled movements called dyskinesias. A drug called amantadine can reduce these movements. To date, there are no objective measures of these movements. The purpose of this study is to measure the reduction of the movements by amantadine and/or topiramate using an objective measure.

DETAILED DESCRIPTION:
Nearly all Parkinson's disease (PD) patients eventually develop abnormal and unwanted movements (dyskinesias) caused by the gold standard treatment, Levodopa. The severity of these movements can range from subtle to extremely debilitating and may or may not interfere with normal activities such as putting on a coat or brushing ones teeth. Currently, one of the very few treatments for these unwanted and involuntary movements is Amantadine. New options to treat dyskinesia would be clinically very valuable. In a previous study, we developed an objective measuring device to quantify dyskinesia.

All PD participants will receive all three of the drug treatment intervention (placebo, Amantadine 300 mg, Amantadine 300 mg plus Topiramate 150 mg). After 2 weeks of one drug treatment, the participants will complete an overnight visit at the OCTRI Inpatient unit. During the next day, participants will complete a mental task while standing on a force plate for one minute every half hour until the end of the study. A levodopa IV infusion will occur from 0900 to 1100. The subjects will be split into 'high' and 'low' dose groups. Those who take <50 mg/hour of oral levodopa or levodopa equivalents will be considered 'low' dose subjects and will receive 1 mg/kg/hr of IV Levodopa during the study visits (1, 2, and 3). Those who administer > 50 mg/hr of oral levodopa to themselves normally will be considered 'high' dose subjects and will received 1.5 mg/kg/hr levodopa. Both groups will receive the infusion for two hours from 0900 - 1100. The study drug will be taken orally at 0800.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease
* At least 21 years of age
* Must be taking Oral levodopa
* Must have dyskinesias by history or previous clinical observation

Exclusion Criteria:

* Significant cognitive impairment as measured by the Montreal Cognitive Assessment (MOCA) score of < 25
* Subjects with unstable medical or psychiatric conditions (including hallucinations)
* Use of dopamine receptor blocking medications (e.g., neuroleptics, certain antiemetics, tetrabenazine)
* History of unstable medical conditions (ie active cardiovascular disease, recent unwellness or surgery etc.)
* Use of anticoagulants
* Current substance abuse
* Previous adverse event on amantadine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Chung, MD, Principal Investigator — Oregon Health & Science University, Portland VA Medical Center; John G Nutt, MD, Principal Investigator — Oregon Health & Science Unversity
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snow BJ, Macdonald L, Mcauley D, Wallis W. The effect of amantadine on levodopa-induced dyskinesias in Parkinson's disease: a double-blind, placebo-controlled study. Clin Neuropharmacol. 2000 Mar-Apr;23(2):82-5. doi: 10.1097/00002826-200003000-00004. PMID 10803797
- [Background] Verhagen Metman L, Del Dotto P, van den Munckhof P, Fang J, Mouradian MM, Chase TN. Amantadine as treatment for dyskinesias and motor fluctuations in Parkinson's disease. Neurology. 1998 May;50(5):1323-6. doi: 10.1212/wnl.50.5.1323. PMID 9595981
- [Background] Del Dotto P, Pavese N, Gambaccini G, Bernardini S, Metman LV, Chase TN, Bonuccelli U. Intravenous amantadine improves levadopa-induced dyskinesias: an acute double-blind placebo-controlled study. Mov Disord. 2001 May;16(3):515-20. doi: 10.1002/mds.1112. PMID 11391748
- [Background] Hagell P, Widner H. Clinical rating of dyskinesias in Parkinson's disease: use and reliability of a new rating scale. Mov Disord. 1999 May;14(3):448-55. doi: 10.1002/1531-8257(199905)14:33.0.co;2-0. PMID 10348468
- [Background] da Silva-Junior FP, Braga-Neto P, Sueli Monte F, de Bruin VM. Amantadine reduces the duration of levodopa-induced dyskinesia: a randomized, double-blind, placebo-controlled study. Parkinsonism Relat Disord. 2005 Nov;11(7):449-52. doi: 10.1016/j.parkreldis.2005.05.008. Epub 2005 Sep 9. PMID 16154788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 individuals were screened for this study. 3 participants were enrolled in the study. 1 participant screen failed due to inability to reduce/stop Amantadine.
Groups:
- Amantadine, Then Amantadine + Topiramate, Then Placebo: Amantadine: Amantadine 200 mg capsule two times a day (week 1); Amantadine 300 mg capsule three times a day (week 2) then 7 Days washout then Amantadine +Topiramate: Amantadine, 200 mg capsule, two times a day with Topiramate 25 mg capsule two times a day (week 1), then Amantadine 300 mg capsule three times a day with Topiramate 50 mg capsule two times a day (week 2) then 7 Days washout then Placebo: Sugar pill 2 capsule three times a day, 2 weeks
- Amantadine + Topiramate, Then Placebo, Then Amantadine: Amantadine +Topiramate: Amantadine, 200 mg capsule, two times a day with Topiramate 25 mg capsule two times a day (week 1), then Amantadine 300 mg capsule three times a day with Topiramate 50 mg capsule two times a day (week 2) then 7 Days washout then Placebo: Sugar pill 2 capsule three times a day, 2 weeks then 7 Days washout then Amantadine: Amantadine 200 mg capsule two times a day (week 1); Amantadine 300 mg capsule three times a day (week 2)
- Placebo, Then Amantadine, Then Amantadine + Topiramate: Placebo: Sugar pill 2 capsule three times a day, 2 weeks then 7 Days washout then Amantadine: Amantadine 200 mg capsule two times a day (week 1); Amantadine 300 mg capsule three times a day (week 2) then 7 Days washout then Amantadine +Topiramate: Amantadine, 200 mg capsule, two times a day with Topiramate 25 mg capsule two times a day (week 1), then Amantadine 300 mg capsule three times a day with Topiramate 50 mg capsule two times a day (week 2)
Period: Overall Study
Arm/Group | Amantadine, Then Amantadine + Topiramate, Then Placebo | Amantadine + Topiramate, Then Placebo, Then Amantadine | Placebo, Then Amantadine, Then Amantadine + Topiramate
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Amantadine 300 mg : Amantadine, 300 mg, capsule, three times a day, two weeks or Amantadine 300 mg : Amantadine, 300 mg, capsule, three times a day, two weeks
  Topiramate : Topiramate, 25 mg, capsule, two times a day, 1 week Sugar Pill, capsule, one time a day, 1 week Topiramate, 50 mg, capsule, three times a day, 1 week or Sugar Pill : sugar pill, capsule, three times a day, 2 weeks
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3
MoCA total [Mean (Standard Deviation); unit: units on a scale] — The MoCA is a short cognitive screening test designed to assist health care professionals for the detection of mild cognitive impairment. The MoCA assesses cognitive function across a variety of domains. The MoCA is scored on a 0 to 30 scale, with lower numbers indicating more cognitive impairment. A point is added to the MoCA if the subject's education high school or less (12 years or less education). Scores ranging from 26 - 30 are normal, 18 - 26 mild impairment, 10 - 17 moderate impairment, and less than 10 severe cognitive impairment.
  units on a scale | 27.7 (1.3)
UPDRS (Part III) Total Score [Mean (Standard Deviation); unit: units on a scale] — This is the motor subsection of the UPDRS and is a commonly used tool to rate the symptoms of Parkinson's disease. Each item on the scale is rated from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. Total score ranges from 0 to 108 with higher values on this scale represent a more severe stage of the disease.
  units on a scale | 16.0 (1.0)
mAIMS [Mean (Standard Deviation); unit: units on a scale] — Modified Abnormal Involuntary Movment Rating Scale (mAIMS) is a commonly utilized scale that is completed by an observer who judges the severity of dyskinesia in 7 body parts (face, neck, trunk, both legs, and both arms). All body parts are rated separately on this 0 (none) to 4 (severe - markedly impairs activities) scale. Thus, the total score can range from 0 - 28 with 28 indicating severe dyskinesia.
  units on a scale | 7 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Forceplate AUC
Description: Area under the curve for the root mean squared velocity in the anterior-posterior direction as measured by a forceplate.
Time Frame: Every 1/2 hour for 8 hour levodopa cycle
Population: triple cross-over study design.
Measure: Mean (Standard Deviation); unit: (meters/second)*hours
Groups:
- Amantadine: Amantadine 300 mg : Amantadine, 300 mg, capsule, three times a day, two weeks
- Amantadine Plus Topiramate: Amantadine 300 mg : Amantadine, 300 mg, capsule, three times a day, two weeks
  Topiramate : Topiramate, 25 mg, capsule, two times a day, 1 week Sugar Pill, capsule, one time a day, 1 week Topiramate, 50 mg, capsule, three times a day, 1 week
- Sugar Pill: Sugar Pill : sugar pill, capsule, three times a day, 2 weeks
Arm/Group | Amantadine | Amantadine Plus Topiramate | Sugar Pill
Number analyzed (Participants) | 3 | 3 | 3
(meters/second)*hours | 10.4 (5.6) | 9.4 (3.5) | 19.1 (18.8)

2. Secondary Outcome: Modified Abnormal Involuntary Movement Scale Area Under the Curve
Description: Area under the curve computed for whole body (total) mAIMS (Modified Abnormal Involuntary Movement Scale) scores at each time measurement. This is a commonly utilized scale that is completed by an observer who judges the severity of levodopa induced dyskinesia (LID) in 7 body parts (face, neck, trunk, both legs, and both arms). All body parts are rated separately on this 0 (none) to 4 (severe - markedly impairs activities) scale. Thus, the total score can range from 0 - 28 with 28 indicating the most severe LID. mAIMS ratings occur as the subject performs the cognitive task while standing on the force plate. mAIMS ratings are made every half hour during the levodopa (LD) dose cycle.
Time Frame: Measured every 1/2 hour for a levodopa dose cycle (starting 1 hour prior to infusion and ending 4 hours post 2-hour infusion)
Measure: Mean (Standard Deviation); unit: Units on a Scale * Hours
Arm/Group | Amantadine | Amantadine Plus Topiramate | Sugar Pill
Number analyzed (Participants) | 3 | 3 | 3
Units on a Scale * Hours | 4.0 (2.9) | 5.3 (4.4) | 8.5 (8.6)

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Amantadine | Amantadine Plus Topiramate | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine (N=3) | Amantadine Plus Topiramate (N=3) | Sugar Pill (N=3)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HALLUCINATIONS (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 0 (0) | 1 (1)
PARESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes